CLINICAL TRIAL: NCT03667638
Title: The Influence of Autologous Platelet Concentrates on Human Keratinocyte Proliferation in Vitro and Wound Healing in Vivo
Brief Title: Influence of Platelet Concentrates on Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Paulmann, Anastasia, Principal Investigator, Hannover Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #1055-2011
Record Dates: First submitted 2018-09-09; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Platelet-Rich Plasma; Wound Healing Delayed
Keywords: Platelet-Rich Plasma; Laser Doppler Imaging; Growth Factors; Wound Healing; Chronic wound healing disorder; Wound quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP Intervention (Experimental): PRP injection into wound border
  Interventions: Combination Product: Platelet-Rich Plasma

INTERVENTIONS:
Combination Product: Platelet-Rich Plasma — Adding PRP to wound bed during surgical debridement
  Other Names: PRP, PMC

SUMMARY:
Chronic soft tissues defects can extend into the fat layer or even deeper and can cause functional disadvantages. Split-thickness skin grafts (STSGs) used to cover these wounds have varying success rates. To improve wound healing in chronic wounds the authors have studied the application of autologous platelet concentrates in a human keratinocyte culture model in vitro and in a combination with surgical procedures in vivo as second line therapy in patients with initially failed wound closure.

DETAILED DESCRIPTION:
For in vitro testing on keratinocytes a platelet-mediator concentrate (PMC) was processed with a commercially available bed-side system (ATR®, Curasan, Germany). In a clinical study soft tissue defects (n=5) were treated using a combination of surgical debridement and autologous platelet rich plasma (PRP). Time of healing as determined by epithelization as well as Laser Doppler Imaging to visualize blood flow were analyzed. Additionally, changes in "ease of surgical wound closure" were determined. Finally, the quality of life of patients was assessed using a validated questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* exposed tendons, ligaments or bone for >3 weeks
* no healing tendency

Exclusion Criteria:

* sepsis
* intensive care treatment
* continuous smoking
* pregnancy or breast feeding women
* participants of other studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Wound Closure | 4 weeks
  Area of wound closure in % compared to initial size

SECONDARY OUTCOMES:
Blood Flow | 4 weeks
  Blood flow measured in wound margins and wound bed compared to regular skin measured using Laser Doppler Imaging
Wound Quality of Life | 21 days
  Quality of patients' life measured using Wound-QoL® Questionnaire before and after Intervention. Seventeen items are included in the Wound-QoL, which could be attributed to three subscales on everyday life, body, and psyche. The paper presents the overall score. A higher value correlates with more wound related burden, meaning a lower value indicates higher qulitiy of life.
  More information: https://www.ncbi.nlm.nih.gov/pubmed/24899053
Ease of surgical wound closure | 21 days
  Estimated ease of surgical wound closure. The patients'wound was discussed by at least two surgeons to obtain agreement on a 14- point "Ease of Closure" scale. This was done on day 0 as well as day 21. The scale ranged from a score of 0, meaning the wound was closed or so small as to require no closure technique, to a score of 13, meaning that it was not possible to close the wound with known reconstructive surgical techniques. A higher value therefore correlates with more complex surgery.
  More information: https://www.ncbi.nlm.nih.gov/pubmed/10231510

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vogt, MD, Principal Investigator — Medical School Hannover
Locations (1):
- Medical School Hannover, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Danielsen P, Jorgensen B, Karlsmark T, Jorgensen LN, Agren MS. Effect of topical autologous platelet-rich fibrin versus no intervention on epithelialization of donor sites and meshed split-thickness skin autografts: a randomized clinical trial. Plast Reconstr Surg. 2008 Nov;122(5):1431-1440. doi: 10.1097/PRS.0b013e318188202c. PMID 18971727
- [Background] Gould L, Abadir P, Brem H, Carter M, Conner-Kerr T, Davidson J, DiPietro L, Falanga V, Fife C, Gardner S, Grice E, Harmon J, Hazzard WR, High KP, Houghton P, Jacobson N, Kirsner RS, Kovacs EJ, Margolis D, McFarland Horne F, Reed MJ, Sullivan DH, Thom S, Tomic-Canic M, Walston J, Whitney JA, Williams J, Zieman S, Schmader K. Chronic wound repair and healing in older adults: current status and future research. J Am Geriatr Soc. 2015 Mar;63(3):427-38. doi: 10.1111/jgs.13332. Epub 2015 Mar 6. PMID 25753048
- [Background] Asadi M, Alamdari DH, Rahimi HR, Aliakbarian M, Jangjoo A, Abdollahi A, Bahar MM, Azadmand A, Forghani N, Sadegh MN, Khayamy ME, Seifalian A. Treatment of life-threatening wounds with a combination of allogenic platelet-rich plasma, fibrin glue and collagen matrix, and a literature review. Exp Ther Med. 2014 Aug;8(2):423-429. doi: 10.3892/etm.2014.1747. Epub 2014 May 29. PMID 25009595
- [Background] Behm B, Babilas P, Landthaler M, Schreml S. Cytokines, chemokines and growth factors in wound healing. J Eur Acad Dermatol Venereol. 2012 Jul;26(7):812-20. doi: 10.1111/j.1468-3083.2011.04415.x. Epub 2011 Dec 26. PMID 22211801
- [Background] Alsousou J, Thompson M, Hulley P, Noble A, Willett K. The biology of platelet-rich plasma and its application in trauma and orthopaedic surgery: a review of the literature. J Bone Joint Surg Br. 2009 Aug;91(8):987-96. doi: 10.1302/0301-620X.91B8.22546. PMID 19651823
- [Background] Werner S, Grose R. Regulation of wound healing by growth factors and cytokines. Physiol Rev. 2003 Jul;83(3):835-70. doi: 10.1152/physrev.2003.83.3.835. PMID 12843410
- [Background] Carter CA, Jolly DG, Worden CE Sr, Hendren DG, Kane CJ. Platelet-rich plasma gel promotes differentiation and regeneration during equine wound healing. Exp Mol Pathol. 2003 Jun;74(3):244-55. doi: 10.1016/s0014-4800(03)00017-0. PMID 12782011
- [Background] Achora S, Muliira JK, Thanka AN. Strategies to promote healing of split thickness skin grafts: an integrative review. J Wound Ostomy Continence Nurs. 2014 Jul-Aug;41(4):335-9; quiz E1-2. doi: 10.1097/WON.0000000000000035. PMID 24988511
- [Background] Appel TR, Potzsch B, Muller J, von Lindern JJ, Berge SJ, Reich RH. Comparison of three different preparations of platelet concentrates for growth factor enrichment. Clin Oral Implants Res. 2002 Oct;13(5):522-8. doi: 10.1034/j.1600-0501.2002.130512.x. PMID 12453130
- [Background] Cohn CS, Lockhart E. Autologous platelet-rich plasma: evidence for clinical use. Curr Opin Hematol. 2015 Nov;22(6):527-32. doi: 10.1097/MOH.0000000000000183. PMID 26390166
- [Background] Berg L, Meyer S, Ipaktchi R, Vogt PM, Muller A, de Zwaan M. [Psychosocial Distress at Different Time Intervals after Burn Injury]. Psychother Psychosom Med Psychol. 2017 Jun;67(6):231-239. doi: 10.1055/s-0042-111006. Epub 2016 Sep 29. German. PMID 27685256
- [Background] House SL. Psychological distress and its impact on wound healing: an integrative review. J Wound Ostomy Continence Nurs. 2015 Jan-Feb;42(1):38-41. doi: 10.1097/WON.0000000000000080. PMID 25549307
- [Background] Blome C, Baade K, Debus ES, Price P, Augustin M. The "Wound-QoL": a short questionnaire measuring quality of life in patients with chronic wounds based on three established disease-specific instruments. Wound Repair Regen. 2014 Jul-Aug;22(4):504-14. doi: 10.1111/wrr.12193. PMID 24899053
- [Background] Weibrich G, Kleis WK. Curasan PRP kit vs. PCCS PRP system. Collection efficiency and platelet counts of two different methods for the preparation of platelet-rich plasma. Clin Oral Implants Res. 2002 Aug;13(4):437-43. doi: 10.1034/j.1600-0501.2002.130413.x. PMID 12175382
- [Background] Weibrich G, Kleis WK, Hafner G, Hitzler WE, Wagner W. Comparison of platelet, leukocyte, and growth factor levels in point-of-care platelet-enriched plasma, prepared using a modified Curasan kit, with preparations received from a local blood bank. Clin Oral Implants Res. 2003 Jun;14(3):357-62. doi: 10.1034/j.1600-0501.2003.00810.x. PMID 12755786
- [Background] Okuda K, Kawase T, Momose M, Murata M, Saito Y, Suzuki H, Wolff LF, Yoshie H. Platelet-rich plasma contains high levels of platelet-derived growth factor and transforming growth factor-beta and modulates the proliferation of periodontally related cells in vitro. J Periodontol. 2003 Jun;74(6):849-57. doi: 10.1902/jop.2003.74.6.849. PMID 12886996
- [Background] Kawase T. Platelet-rich plasma and its derivatives as promising bioactive materials for regenerative medicine: basic principles and concepts underlying recent advances. Odontology. 2015 May;103(2):126-35. doi: 10.1007/s10266-015-0209-2. Epub 2015 Jun 4. PMID 26040505
- [Background] Amable PR, Carias RB, Teixeira MV, da Cruz Pacheco I, Correa do Amaral RJ, Granjeiro JM, Borojevic R. Platelet-rich plasma preparation for regenerative medicine: optimization and quantification of cytokines and growth factors. Stem Cell Res Ther. 2013 Jun 7;4(3):67. doi: 10.1186/scrt218. PMID 23759113
- [Background] Nurden AT, Nurden P, Sanchez M, Andia I, Anitua E. Platelets and wound healing. Front Biosci. 2008 May 1;13:3532-48. doi: 10.2741/2947. PMID 18508453
- [Background] Barrientos S, Stojadinovic O, Golinko MS, Brem H, Tomic-Canic M. Growth factors and cytokines in wound healing. Wound Repair Regen. 2008 Sep-Oct;16(5):585-601. doi: 10.1111/j.1524-475X.2008.00410.x. PMID 19128254
- [Background] Cho JW, Kim SA, Lee KS. Platelet-rich plasma induces increased expression of G1 cell cycle regulators, type I collagen, and matrix metalloproteinase-1 in human skin fibroblasts. Int J Mol Med. 2012 Jan;29(1):32-6. doi: 10.3892/ijmm.2011.803. Epub 2011 Sep 30. PMID 21964487
- [Background] Carmeliet P, Jain RK. Molecular mechanisms and clinical applications of angiogenesis. Nature. 2011 May 19;473(7347):298-307. doi: 10.1038/nature10144. PMID 21593862
- [Background] Mammoto T, Jiang A, Jiang E, Mammoto A. Platelet rich plasma extract promotes angiogenesis through the angiopoietin1-Tie2 pathway. Microvasc Res. 2013 Sep;89:15-24. doi: 10.1016/j.mvr.2013.04.008. Epub 2013 May 6. PMID 23660186
- [Background] Burnouf T, Tseng YH, Kuo YP, Su CY. Solvent/detergent treatment of platelet concentrates enhances the release of growth factors. Transfusion. 2008 Jun;48(6):1090-8. doi: 10.1111/j.1537-2995.2008.01691.x. Epub 2008 Mar 25. PMID 18373502
- [Background] Shaw TJ, Martin P. Wound repair at a glance. J Cell Sci. 2009 Sep 15;122(Pt 18):3209-13. doi: 10.1242/jcs.031187. No abstract available. PMID 19726630
- [Background] Eppley BL, Woodell JE, Higgins J. Platelet quantification and growth factor analysis from platelet-rich plasma: implications for wound healing. Plast Reconstr Surg. 2004 Nov;114(6):1502-8. doi: 10.1097/01.prs.0000138251.07040.51. PMID 15509939
- [Background] Kaltalioglu K, Coskun-Cevher S. A bioactive molecule in a complex wound healing process: platelet-derived growth factor. Int J Dermatol. 2015 Aug;54(8):972-7. doi: 10.1111/ijd.12731. Epub 2014 Oct 14. PMID 25312059
- [Background] Anitua E, Aguirre JJ, Algorta J, Ayerdi E, Cabezas AI, Orive G, Andia I. Effectiveness of autologous preparation rich in growth factors for the treatment of chronic cutaneous ulcers. J Biomed Mater Res B Appl Biomater. 2008 Feb;84(2):415-21. doi: 10.1002/jbm.b.30886. PMID 17595032
- [Background] Martinez-Zapata MJ, Marti-Carvajal AJ, Sola I, Exposito JA, Bolibar I, Rodriguez L, Garcia J. Autologous platelet-rich plasma for treating chronic wounds. Cochrane Database Syst Rev. 2012 Oct 17;10:CD006899. doi: 10.1002/14651858.CD006899.pub2. PMID 23076929
- [Background] Kim SA, Ryu HW, Lee KS, Cho JW. Application of platelet-rich plasma accelerates the wound healing process in acute and chronic ulcers through rapid migration and upregulation of cyclin A and CDK4 in HaCaT cells. Mol Med Rep. 2013 Feb;7(2):476-80. doi: 10.3892/mmr.2012.1230. Epub 2012 Dec 12. PMID 23242428
- [Background] Reinke JM, Sorg H. Wound repair and regeneration. Eur Surg Res. 2012;49(1):35-43. doi: 10.1159/000339613. Epub 2012 Jul 11. PMID 22797712
- [Background] Mazzucco L, Borzini P, Gope R. Platelet-derived factors involved in tissue repair-from signal to function. Transfus Med Rev. 2010 Jul;24(3):218-34. doi: 10.1016/j.tmrv.2010.03.004. PMID 20656189
- [Background] Robson MC, Maggi SP, Smith PD, Wassermann RJ, Mosiello GC, Hill DP, Cooper DM. Original articles: ease of wound closure as an endpoint of treatment efficacy. Wound Repair Regen. 1999 Mar-Apr;7(2):90-6. doi: 10.1046/j.1524-475x.1999.00090.x. PMID 10231510
- [Background] Limbourg A, Korff T, Napp LC, Schaper W, Drexler H, Limbourg FP. Evaluation of postnatal arteriogenesis and angiogenesis in a mouse model of hind-limb ischemia. Nat Protoc. 2009;4(12):1737-46. doi: 10.1038/nprot.2009.185. Epub 2009 Nov 5. PMID 19893509
- [Background] Khatib M, Jabir S, Fitzgerald O'Connor E, Philp B. A systematic review of the evolution of laser Doppler techniques in burn depth assessment. Plast Surg Int. 2014;2014:621792. doi: 10.1155/2014/621792. Epub 2014 Aug 7. PMID 25180087
- [Background] Paul DW, Ghassemi P, Ramella-Roman JC, Prindeze NJ, Moffatt LT, Alkhalil A, Shupp JW. Noninvasive imaging technologies for cutaneous wound assessment: A review. Wound Repair Regen. 2015 Mar-Apr;23(2):149-62. doi: 10.1111/wrr.12262. PMID 25832563
- [Background] Xian LJ, Chowdhury SR, Bin Saim A, Idrus RB. Concentration-dependent effect of platelet-rich plasma on keratinocyte and fibroblast wound healing. Cytotherapy. 2015 Mar;17(3):293-300. doi: 10.1016/j.jcyt.2014.10.005. Epub 2014 Nov 21. PMID 25456581
- [Background] Gilliver SC, Ashworth JJ, Ashcroft GS. The hormonal regulation of cutaneous wound healing. Clin Dermatol. 2007 Jan-Feb;25(1):56-62. doi: 10.1016/j.clindermatol.2006.09.012. PMID 17276202
- [Derived] Paulmann A, Strauss S, Limbourg A, Vogt PM. Platelet-derived concentrates influence human keratinocyte proliferation in vitro and induce wound healing in a prospective case series of chronic wounds of different entities in vivo. Innov Surg Sci. 2022 Oct 10;7(2):45-58. doi: 10.1515/iss-2022-0011. eCollection 2022 Jun. PMID 36317012